CLINICAL TRIAL: NCT04925583
Title: Magnetic Resonance Guided Adaptive Stereotactic Body Radiotherapy for Lung Tumors in Ultracentral Location
Acronym: MAGELLAN
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Department Head, University Hospital Heidelberg
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RADONK-Magellan_2020
Record Dates: First submitted 2021-05-18; First posted 2021-06-14 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer
Keywords: SBRT; IGRT; MR-guidance; ultracentral lung tumor; NSCLC; oligometastases
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Dose escalation, Arm 1: Level 0, 5.0 Gy, 10 fractions Arm 2: Level 1, 5.5 Gy, 10 fractions Arm 3: Level 2, 6.0 Gy, 10 fractions Arm 4: Level 3, 6.5 Gy, 10 fractoins
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Level 0 (Experimental): Total dose 50 Gy, (10 x 5 Gy single dose)
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT)
- Level 1 (Experimental): Total dose 55 Gy, (10 x 5.5 Gy single dose)
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT)
- Level 2 (Experimental): Total dose 60 Gy, (10 x 6 Gy single dose)
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT)
- Level 3 (Experimental): Total dose 65 Gy, (10 x 6.5 Gy single dose)
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy (SBRT) — * level 0 (de-escalation): 10 x 5.0Gy
  * level 1 (start): 10 x 5.5Gy
  * level 2: 10 x 6.0Gy
  * level 3: 10 x 6.5Gy

SUMMARY:
MAGELLAN is a phase-I dose escalation trial that aims to identify the maximum tolerated dose (MTD) of MR-guided SBRT of ultracentral lung Tumors (primary objective). Thus, a maximum of 38 patients with ultracentral lung tumors (overlap of the planning target volume with the proximal bronchial tree and/or esophagus) will receive MR-guided SBRT including gated dose delivery and daily plan adaptation on a 0.35 MR-linac System. Dose levels are as follows:

* 0 (de-escalation): 10 x 5.0Gy
* 1 (start): 10 x 5.5Gy
* 2: 10 x 6.0Gy
* 3: 10 x 6.5Gy

Dose escalation is performed according to a time-to-event continual reassessment method (TITE-CRM) with backup element. Patients are observed individually for 12 months to detect potential dose limiting toxicity (DLT = primary endpoint) and for a total of 24 months to detect potential tumor relapse.

DETAILED DESCRIPTION:
Stereotactic body radiotherapy (SBRT) is a well-established local treatment method for early-stage NSCLC or lung metastases. However, clinicians are restricted in the utilization of sufficiently high radiation doses when the lung tumor is in ultracentral location next to radiosensitive organs-at-risk (OAR, e.g. the central airways or the esophagus). MR-guided SBRT can minimize the dose to these OAR by advanced techniques to correct for interfractional (daily plan adaptation) and intrafractional motion (respiratory gating, i.e. synchronization of beam delivery to the patient's breathing). Consequently, the MAGELLAN trial uses MR-guided SBRT to enable safe dose escalation to ultracentral lung tumors. The primary objective of this phase I dose escalation trial is to detect the maximum tolerated dose of MR-guided SBRT to ultracentral lung tumors with a dose limiting toxicity (DLT) rate = 35%. This dose should yield the optimum balance between acceptable treatment toxicity and good tumor control. The corresponding primary endpoint is the observation of the binary outcome dose-limiting toxicity (DLT) within 12 months from start of radiation. Secondary objectives include description of tumor control, patient survival and patient-reported outcomes, assessment of longitudinal cardiopulmonary function and dosimetry evaluations. Exploratory objectives include detection of early biomarkers of pulmonary toxicity and tumor response from multiparamtetric thoracic MRI examinations as well as peripheral blood samples before and early after treatment. A maximum of 38 adult patients may be accrued. Inclusion criteria encompass indication for pulmonary SBRT, ultracentral lung tumor location defined as overlap of the planning target volume (PTV) with the proximal bronchial tree or esophagus and a maximum tumor diameter ≤ 5cm. MR-guided SBRT is delivered on a 0.35T MR-Linac (6MV linear accelerator) with daily plan adaptation and gated dose delivery. Four dose levels may be employed:

* 0 (de-escalation): 10 x 5.0Gy
* 1 (start): 10 x 5.5Gy
* 2: 10 x 6.0Gy
* 3: 10 x 6.5Gy

Dose level 0 represents a de-escalation step which is deemed safe by retrospective clinical data. Dose level 3 confidently reaches a BED10 > 100 Gy necessary for adequate local tumor control in the lung according to hitherto data. Individual observation time for DLTs is 12 months. Dose escalation is performed in dose escalation cohorts consisting of three patients (N = 3) and the first cohort starts at dose level 1 (10 x 5.5 Gy). A time-to-event continual reassessment method (TITE-CRM) is used to recommend the dose level for the next cohort after a cumulative observation time of 18 months. TITE-CRM accounts for all available data at any given time to estimate DLT rates for each dose level and will recommend the dose level closest to the MTD. Admissible patients who present during the cumulative observation time are included as backup patients and treated on the dose level below the current recommendation. An escalation with overdose control (EWOC) approach is applied to prevent treatment with too toxic doses. According to the stopping criteria, patient accrual will be stopped after including 36 patients or 40 months after the first subject in date (recruitment of current dose escalation cohort may be completed), in case that estimation of the MTD is sufficiently certain or if all dose levels appear too toxic. After patient accrual has been stopped and all patients have completed their individual observation time, a final dose recommendaton will be performed which represents the MTD estimate. During follow-up, patients receive clinical assessments (3 monthly), thoracic CT- (3-monthly) and MR-imaging (after 3 months), one cardiology assessment (after 12 months), pulmonary function testing (12-monthly) and peripheral blood samples (last treatment day, after 3 months) for a total of 2 years after treatment.

ELIGIBILITY:
Inclusion Criteria:

* ultracentral location of the lung tumor, which is defined as an expected contact or overlap of the planning target volume with the proximal bronchial tree or esophagus at the time of consultation
* indication for SBRT of the ultracentral pulmonary tumor
* maximum diameter of the ultracentral pulmonary tumor < 5cm
* age > 18 years of age
* Karnofsky Performance Score > 70% (ECOG Score 0 - 2)
* ability to lie still on the MR-linac table for at least one hour
* ability to hold one's breath for more than 20 seconds
* successful completion of MRgRT simulation
* for women with childbearing potential, adequate contraception.
* ability of subject to understand character and individual consequences of the clinical trial
* written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

* refusal of the patients to take part in the study
* previous radiotherapy of the lung and mediastinum, if previous and current target volumes overlap
* patients who have not yet recovered from acute toxicities of prior therapies
* (planned) treatment with vascular endothelial growth factor (VEGF) inhibitors, e.g. Bevacizumab, within the time interval 2 weeks before and 2 weeks after SBRT
* pregnant or lactating women
* contraindications against performing MRI scans (pacemakers, other implants making MRI impossible)
* participation in another competing clinical study or observation period of competing trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | For 12 months from the beginning of SBRT.
  Observation of the binary outcome dose-limiting toxicity (DLT). DLTs are defined in a catalogue of mainly pulmonary, esophageal and cardiac toxicity based on the CTCAE in Version 5.0.

SECONDARY OUTCOMES:
Local tumor control | For 24 months upon enrollment
  Total number of treated ultracentral tumor.
Regional tumor control | For 24 months upon enrollment
  Number of tumor leasions in Lungs and Mediastinum excluding the treated ultracentral tumor.
Distant tumor Control | For 24 months upon enrollment
  Number of Tumor leasions Outside lungs and mediastinum.
Progression-free survival | For 24 months upon enrollment
Overall survival | For 24 months upon enrollment
EORTC QLQ C-30 | For 24 months upon enrollment
  Changes in quality of life following MR-guided ultracentral lung SBRT, according to EORTC QLQ C-30.
EORTC QLQ-LC13 | For 24 months upon enrollment
  Changes in quality of life following MR-guided ultracentral lung SBRT, according to EORTC QLQ-LC13.
Vital Capacity | For 24 months upon enrollment
  Pulmonary function test parameter.
Forced Expiratory Volume in the 1st second | For 24 months upon enrollment
  Pulmonary function test parameter.
Cardiovascular function: Longitudinal strain | For 12 months upon enrollment
  Echocardiography.
Cardiovascular function: Left ventricular ejection fraction (LVEF) | For 12 months upon enrollment
  Echocardiography.
Cardiovascular function: Ratio between early mitral inflow velocity and mitral annular early diastolic velocity (E/e') | For 12 months upon enrollment
  Echocardiography.
Cardiovascular function: N-terminal prohormone of brain natriuretic peptide (NT-proBNP) | For 12 months upon enrollment
  Blood Sample.
Cardiovascular function: High-sensitive Troponin-T (hsTNT) | For 12 months upon enrollment
  Blood Sample.
Dosimetry parameters of MRgRT as compared to CT-based SBRT techniques | through study completion, an average of 1 year
Apparent Diffusion Coefficient (ADC) | 3 months upon SBRT.
  Translational imaging biomarkers based on multiparametric MRI (T1w, T2w and diffusion-weighted) for early detection of pulmonary toxicity and tumor relapse (explorative).
Serum cytokines | Immediately and 3 months upon SBRT.
  Translational blood biomarkers (explorative).
Immunophenotypes of peripheral blood mononucleated cells (PBMC) | Immediately and 3 months upon SBRT.
  Translational blood biomarkers for early detection of pulmonary toxicity and tumor relapse (explorative).

CONTACTS AND LOCATIONS:
Overall Officials: Juliane Hörner-Rieber, PD, Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hospital of Heidelberg, Radiation Oncology, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Regnery S, Ristau J, Weykamp F, Hoegen P, Sprengel SD, Paul KM, Buchele C, Kluter S, Rippke C, Renkamp CK, Pohl M, Meis J, Welzel T, Adeberg S, Koerber SA, Debus J, Horner-Rieber J. Magnetic resonance guided adaptive stereotactic body radiotherapy for lung tumors in ultracentral location: the MAGELLAN trial (ARO 2021-3). Radiat Oncol. 2022 May 25;17(1):102. doi: 10.1186/s13014-022-02070-x. PMID 35614486